CLINICAL TRIAL: NCT03170752
Title: Implementing and Testing a Cardiovascular Assessment Screening Program to Promote Healthy Aging (CASP)
Brief Title: Implementing and Testing a Cardiovascular Assessment Screening Program (CASP)
Acronym: CASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Jill Bruneau, Doctoral candidate, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 20180318
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Risk Factor; Smoking; Diabetes Mellitus; Dyslipidemias; Hypertension; Physical Activity; Stress, Psychological
Keywords: RCT, Cardiovascular Risk Factors, Screening
MeSH Terms: conditions — Smoking; Diabetes Mellitus; Dyslipidemias; Hypertension; Motor Activity; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The screening intervention Cardiovascular Assessment Screening Program (CASP) to be implemented by NPs in the intervention group has three steps:
  1. Identification of patients (using Eligibility for Heart Health Screening Form, Heart Health Assessment Pamphlet, Tracking Form for Heart Health Screening, Algorithm for NP to Screen);
  2. Screening utilizing appropriate tools (Cardiovascular Screening Checklist, Heart Health Screening Website/App);
  3. Actions to follow up on the screening results (Heart Health Screening Website/App, CV Decision Tree Algorithm).
  Interventions: Behavioral: Cardiovascular Assessment Screening Program (CASP)
- Control group (No Intervention): The NPs in the control group will be instructed to follow usual practice to screen patients for cardiovascular disease.

INTERVENTIONS:
Behavioral: Cardiovascular Assessment Screening Program (CASP) — Step 1. Identification of patients; Step 2. Screening utilizing appropriate tools; and Step 3. Actions to follow up on the screening results.
  Arms: Intervention group

SUMMARY:
This study is a randomized controlled trial (RCT) and there will be two groups: an intervention group and a control group. Nurse practitioners (NPs) across Newfoundland and Labrador (NL) who agree to participate will be randomly assigned to one of the two groups. The NPs in the intervention group will be asked to screen about 30 individuals aged 40-74 years without established cardiovascular disease (CVD) that currently come to their clinics. The NPs will be asked to screen these patients for CVD using a set of specific data collection tools that will be in electronic format. The control group will carry on with usual practice. Their charts will be reviewed by the researchers at a later date. At the end of the study, the screening program, with tools and strategies for CVD screening, will be given to NPs in the control group.

DETAILED DESCRIPTION:
The RCT will be conducted to test the screening intervention, the Cardiovascular Assessment Screening Program, with nurse practitioners across NL.

Research Questions

1. What is the effect of implementing the Cardiovascular Assessment Screening Program on comprehensiveness of screening by nurse practitioners in NL?
2. What is the effect of implementation of the Cardiovascular Assessment Screening Program on the identification of individuals at high risk of CVD within the nurse practitioner practice?
3. What is the effect of implementation of the Cardiovascular Assessment Screening Program on recommendations that are made by nurse practitioners in NL?
4. What components of the Cardiovascular Assessment Screening Program are effective in promoting CVD screening and appropriate follow-up by nurse practitioners in NL?
5. What are the patients' and nurse practitioners' factors that influence participation in the Cardiovascular Assessment Screening Program in NL? The main outcome is the comprehensiveness of CVD screening. The null hypothesis for the RCT is stated as follows: There will be no difference in comprehensiveness of screening between the intervention group and the control group.

Methodology The RCT study will involve implementation and evaluation of the Cardiovascular Assessment Screening Program across the province of NL. The RCT will use block randomization following NP recruitment to allocate participating NP practices to either the intervention group or the control group. The NPs in the intervention group will participate in scheduled face-to-face educational sessions as well as webinars from their workplaces to receive support on using specific tools to identify, screen, and follow-up with patients. The NPs will also receive instructions on data collection methods using the study's Access Database developed by Newfoundland and Labrador Centre for Health Information (NLCHI).

The NPs in the control group will participate in a webinar education session and will be instructed to follow usual practice to screen patients for CVD. The NPs in the control group will receive instructions on keeping a record of patients who were seen in their clinics and whether or not the patients will be eligible to participate in the study based on age and history. This information will be used by researchers to conduct a retrospective chart review on a specified date during the data collection period. The specific CVD screening tools provided to the NPs in the intervention group will be made available to NPs in the control group following conclusion of this study.

Setting & Sample The RCT will take place in community-based clinics with NP practices from both rural and urban areas in the various regional health authorities across NL. NPs may be working in solo practice or working with several other NPs in a group practice. There will be four types of NP practices: 1) rural solo, 2) rural group, 3) urban solo and, 4) urban group. NPs working in the same group practice will need to be allocated to the same group, so block randomization will be used once all of the NP practices have been recruited. Using a random number generator, NP practices will be allocated to either the intervention group or the control group within each block (type) of practice.

The sample size estimation for this study was determined using the proportion of eligible patients who were comprehensively screened as the outcome measure of interest. A study that considered the effectiveness of a national risk assessment program for patients aged 40-74 years found that approximately 40% had complete Health Checks and 60% had partial Health Checks among high risk patients in the United Kingdom (UK) National Health Service Health Check Program (Artec et al., 2013). The sample size for this proposed study was calculated based on the assumption that 40% of the screening will be comprehensive in the control group practices. The research team decided that comprehensive screening of 70% of patients seen by the NPs in the intervention group during this study would indicate an effective intervention. Using a two-sided alpha of 0.05 and 90% power, the sample size was calculated to be 250 patients (125 patients per group). Considering that patients would need to provide consent to participate in this study the research team assumed that 20% of those approached would refuse. This means that 300 patients with 150 patients per group would be required. To be realistic about workload, each NP would need to include 25-30 patients. A minimum of 10 NPs therefore needs to be recruited. The duration of the data collection period will vary by NP according to the number of eligible patients seen. For example, if an NP sees one eligible patient per day for five days a week, then the data collection period would be six weeks for a total of 30 patients. If an NP sees two eligible patients per day, then the data collection period would be three weeks.

ELIGIBILITY:
Inclusion Criteria for NPs:

* Employment as a full-time NP in community-based settings
* Access to healthy, asymptomatic patients between the ages of 40-74 years of age
* Ability of the practice to collect data.

Inclusion Criteria for the Patients:

* Eligible based on age,
* No established CVD (such as coronary heart disease (CHD) or ischemic heart disease (IHD), myocardial infarctions (MIs), congestive heart failure (CHF), transient ischemic attacks (TIAs), cerebrovascular accidents (CVAs), peripheral vascular disease (PVD), and pulmonary emboli (PE).
* Willingness to participate in the study.

Exclusion Criteria

* Age less than 20 or over 75 years
* Established Cardiovascular Disease (such as coronary heart disease (CHD) or ischemic heart disease (IHD), myocardial infarctions (MIs), congestive heart failure (CHF), transient ischemic attacks (TIAs), cerebrovascular accidents (CVAs), peripheral vascular disease (PVD), and pulmonary emboli (PE)).
* Inability to attend NP clinic visit

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-09-29 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are comprehensively screened to the number of eligible patients seen in the intervention group compared to the control group as assessed by the completeness of CV Screening Checklist data collection form. | 6-8 weeks
  If the CV screening Checklist is only partially completed or not completed at all then it will not be considered comprehensive. Logistic regression is used because the outcome is dichotomous (yes or no). The patients had comprehensive screening (Yes) or they did not have comprehensive screening (No).

SECONDARY OUTCOMES:
Identification of individuals at high risk for cardiovascular disease as assessed by the calculated Framingham Risk Score. | 6-8 weeks
  The Framingham Risk Scores of patients in the intervention group will be calculated using an online calculator and the number of high risk individuals will be identified and reported.
The management recommendations that are made by the NPs as assessed by the responses collected on the CV Screening Checklist data collection form (intervention group) and the chart review (control group). | 6-8 weeks
  Chi Square will be used to compare the recommendations made by NPs in the intervention group compared to the NPs in the control group following screening of patients for cardiovascular disease.
The patient and NP factors that influence participation in the CASP as assessed by content analysis of patient and NP feedback questionnaires. | 6-8 weeks
  The responses from the Patient and NP Feedback Questionnaires will be assessed using content analysis to determine the factors that influence participation in the screening intervention Cardiovascular Assessment Screening Program (CASP).

CONTACTS AND LOCATIONS:
Overall Officials: Jill Bruneau, PhD(c), Principal Investigator — Memorial University
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez-Bueno C, Cavero-Redondo I, Martinez-Andres M, Arias-Palencia N, Ramos-Blanes R, Salcedo-Aguilar F. Effectiveness of multifactorial interventions in primary health care settings for primary prevention of cardiovascular disease: A systematic review of systematic reviews. Prev Med. 2015 Jul;76 Suppl:S68-75. doi: 10.1016/j.ypmed.2014.11.028. Epub 2014 Dec 12. PMID 25511466
- [Background] Artac M, Dalton AR, Majeed A, Car J, Millett C. Effectiveness of a national cardiovascular disease risk assessment program (NHS Health Check): results after one year. Prev Med. 2013 Aug;57(2):129-34. doi: 10.1016/j.ypmed.2013.05.002. Epub 2013 May 21. PMID 23701848
- [Background] Avanzini F, Marzona I, Baviera M, Barlera S, Milani V, Caimi V, Longoni P, Tombesi M, Silletta MG, Tognoni G, Roncaglioni MC; Risk and Prevention Study Collaborative Group. Improving cardiovascular prevention in general practice: Results of a comprehensive personalized strategy in subjects at high risk. Eur J Prev Cardiol. 2016 Jun;23(9):947-55. doi: 10.1177/2047487315613664. Epub 2015 Nov 2. PMID 26525065
- [Background] Brindle P, Beswick A, Fahey T, Ebrahim S. Accuracy and impact of risk assessment in the primary prevention of cardiovascular disease: a systematic review. Heart. 2006 Dec;92(12):1752-9. doi: 10.1136/hrt.2006.087932. Epub 2006 Apr 18. PMID 16621883
- [Background] Cardiometabolic Risk Working Group: Executive Committee; Leiter LA, Fitchett DH, Gilbert RE, Gupta M, Mancini GB, McFarlane PA, Ross R, Teoh H, Verma S, Anand S, Camelon K, Chow CM, Cox JL, Despres JP, Genest J, Harris SB, Lau DC, Lewanczuk R, Liu PP, Lonn EM, McPherson R, Poirier P, Qaadri S, Rabasa-Lhoret R, Rabkin SW, Sharma AM, Steele AW, Stone JA, Tardif JC, Tobe S, Ur E. Identification and management of cardiometabolic risk in Canada: a position paper by the cardiometabolic risk working group (executive summary). Can J Cardiol. 2011 Mar-Apr;27(2):124-31. doi: 10.1016/j.cjca.2011.01.016. PMID 21459258
- [Background] Tobe SW, Stone JA, Walker KM, Anderson T, Bhattacharyya O, Cheng AY, Gregoire J, Gubitz G, L'Abbe M, Lau DC, Leiter LA, Oh P, Padwal R, Poirier L, Selby P, Tremblay M, Ward RA, Hua D, Liu PP; C-CHANGE Initiative. Canadian Cardiovascular Harmonized National Guidelines Endeavour (C-CHANGE): 2014 update. CMAJ. 2014 Nov 18;186(17):1299-305. doi: 10.1503/cmaj.140387. Epub 2014 Oct 20. No abstract available. PMID 25332362
- [Derived] Bruneau J, Moralejo D, Parsons K. Evaluating the effectiveness of the cardiovascular assessment screening program with nurse practitioners and patients: results of a cluster randomised controlled trial. BMC Prim Care. 2024 May 24;25(1):185. doi: 10.1186/s12875-024-02432-2. PMID 38789927